CLINICAL TRIAL: NCT00102492
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Fixed-Dose Study Evaluating the Efficacy and Safety of GW679769 in Subjects With Major Depressive Disorder.
Brief Title: Study Of GW679769 In Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKF100092
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Depressive Disorder, Major; Major Depressive Disorder (MDD)
Keywords: Major Depressive Disorder; Major Depression; Mood Disorders; Major Depressive Episode
MeSH Terms: conditions — Depressive Disorder, Major; Mood Disorders | interventions — casopitant

INTERVENTIONS:
Drug: GW679769

SUMMARY:
This is a placebo-controlled, fixed dose study that will evaluate the efficacy and safety of GW679769 in subjects with major depressive disorder.

ELIGIBILITY:
Inclusion criteria:

* Subjects must have the ability to comprehend the key components of the consent form.
* Subject must have met DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision) criteria for current MDE (major depressive episode) for at least 8 weeks prior to the Screening Visit.
* If female, subjects must be practicing an acceptable method of birth control.
* Subjects must have rating scores as outlined.

Exclusion criteria:

* Subjects whose symptoms of the MDE are better accounted for by another diagnosis.
* Subjects with a history of schizophrenia, schizoaffective disorders or bipolar disorder.
* Subjects have a positive urine test for illicit drug use and/or a history of substance abuse or alcohol dependence within the past 12 months.
* Subjects with an unstable medical disorder.
* If female, pregnant or lactating.
* Subjects who have received ECT (electroconvulsive therapy) or TMS (transcranial magnetic stimulation) within the 6 months preceding screening or who have ever been homicidal.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 356 (Actual)
Dates: Start 2004-10; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the 17-item Hamilton Depression Rating Scale (HAM-D) total score at week 8, Last Observation Carried Forward.

SECONDARY OUTCOMES:
CGI, HAM-A, QUIDS, SDS, MOS-12 Sleep Module, LSEQ, Safety and Tolerability, PK/PD

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (26):
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Winter Park, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Smyrna, Georgia
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, Farmington Hills, Michigan
  - GSK Investigational Site, Saint Charles, Missouri
  - GSK Investigational Site, Clementon, New Jersey
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Beachwood, Ohio
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Memphis, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Irving, Texas
  - GSK Investigational Site, Lake Jackson, Texas
  - GSK Investigational Site, Bellevue, Washington
- Canada (4):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Miramichi, New Brunswick
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Sherbrooke, Quebec